CLINICAL TRIAL: NCT00002890
Title: PHASE I DOSE-ESCALATION TRIAL OF YTTRIUM-90-LABELED HuM195 (HUMANIZED ANTI-CD33) IN PATIENTS WITH ADVANCED MYELOID MALIGNANCIES
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Myelodysplastic Syndrome or Relapsed or Refractory Acute Myeloid Leukemia or Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 96-010; CDR0000065213 (Registry Identifier: PDQ (Physician Data Query)); NCI-H96-1100
Record Dates: First submitted 1999-11-01; First posted 2004-08-11 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: recurrent adult acute myeloid leukemia; relapsing chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic | interventions — lintuzumab

INTERVENTIONS:
Biological: lintuzumab

SUMMARY:
RATIONALE: Monoclonal antibodies can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells.

PURPOSE: Phase I trial to study the effectiveness of radiolabeled monoclonal antibody in treating patients with myelodysplastic syndrome or relapsed or refractory acute myeloid leukemia or chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety and toxicity of yttrium-90-labeled humanized monoclonal antibody M195 (90Y-MOAB HuM195) in patients with relapsed or refractory myeloid malignancies. II. Determine the pharmacology and dosimetry of 90Y-MOAB HuM195. III. Study the biological effects of 90Y-MOAB HuM195, including the ability to elicit human anti-human antibody responses and antileukemic responses.

OUTLINE: This study seeks to estimate the maximum tolerated dose (MTD) of yttrium-90-labeled humanized monoclonal antibody M195 (90Y-MOAB HuM195). All patients receive a single intravenous dose of 90Y-MOAB HuM195. Groups of 3 to 6 patients are treated at escalated doses of yttrium-90 until the MTD is determined. Patients with active leukemia who exhibit at least a 50% clearing of marrow blasts after the first dose may receive a second dose after 4-8 weeks provided remaining blasts are CD33-positive, there is no evidence of human anti-human antibody response, and any toxicity has resolved. All patients are followed monthly for 4 months after treatment.

PROJECTED ACCRUAL: Up to 24 patients will be treated. The study is expected to require 12-18 months to complete.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Pathologically confirmed myeloid malignancies as follows: Acute myelogenous leukemia that is relapsed or refractory after at least 2 courses of standard induction chemotherapy Accelerated or myeloblastic chronic myelogenous leukemia Refractory anemia with excess blasts (RAEB) RAEB in transformation Chronic myelomonocytic leukemia More than 25% of bone marrow blasts positive for the CD33 antigen Clear signs of active leukemia following recovery from prior therapy required No rapidly accelerating blast count No clinically unstable disease No active CNS leukemia

PATIENT CHARACTERISTICS: Age: Over 16 Performance status: Karnofsky 60%-100% Life expectancy: At least 6 weeks Hematopoietic: Not specified Hepatic: Bilirubin less than 2.5 mg/dL AST less than 3 times normal Alkaline phosphatase less than 3 times normal Renal: Creatinine less than 2.0 mg/dL Cardiovascular: No NYHA class III/IV status Pulmonary: No clinically significant pulmonary disease Other: No serious infection uncontrolled by antibiotics No pregnant or nursing women Negative pregnancy test required of fertile women

PRIOR CONCURRENT THERAPY: Recovered from prior therapy Biologic therapy: No detectable antibodies to M195 from prior monoclonal antibody M195 or HuM195 Chemotherapy: At least 2 days since hydroxyurea At least 3 weeks since other chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 3 weeks since radiotherapy Surgery: Not specified

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 1996-10; Primary Completion 2001-01 (Actual); Study Completion 2001-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph G. Jurcic, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States